## **PATIENT CONSENT FORM**

Study title: Can an adjustable compression garment replace compression bandaging in the treatment of patients with Breast Cancer related upper limb Lymphoedema? A pilot study

| Yes □ | No □ |
|-------|----------------------------------------|
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No □ |
| Yes □ | No □ |
| | Yes |

| FUTURE CONTACT [please choose one or more as you see fit] | | |
|---|---|---|
| <b>OPTION 1:</b> I consent to be re-contacted by researchers about possible | Yes □ | No □ |
| future research <b>related</b> to the current study for which I may be eligible. | | |
| <b>OPTION 2:</b> I consent to be re-contacted by researchers about possible | | No 🗆 |
| future research <b>unrelated</b> to the current study for which I may be eligible. | | |

Version : 1 Date: 23/10/19 Page 1

| Patient Name (Block Capitals) | | Patient Signature | Date |
|---|---|---|---|
| Translator Name (Block Ca | <br>apitals) | <br>Translator Signature | Date |
| Legal Representative/Gua To be completed by the P | | Legal Representative/Gu | ardian Signature Date |
| purpose of this study in a | way that they o | o fully explain to the above could understand. I have exped them to ask questions or | plained the risks involved as |
| | I | I | I |
| Name (Block Capitals) | Qualificat | ions Signature | Date |

3 copies to be made: 1 for patient, 1 for PI and 1 for hospital records.